CLINICAL TRIAL: NCT03221556
Title: Improving Outcomes for Low-Income Mothers With Depression: A Comparative Effectiveness Trial of Two Brief Interventions in the Patient-Centered Medical Home.
Brief Title: Improving Outcomes for Low-Income Mothers With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: H-36434; AD-1603-34662 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post Partum Depression
Keywords: Comparative effectiveness research; Patient-centered medical home; Shared decision-making
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engagement-Focused Care Coordination (EFCC) (Active Comparator): The brief intervention in Engagement-Focused Care Coordination is the Engagement Interview. In this model, providers meet one to two times with mothers who screen positive for depression, and use techniques of shared decision-making to help mothers process the results of the screen; explore treatment options; and connect with formal mental health services. Engagement-Focused Care Coordination emphasizes referral to formal mental health services.
  Interventions: Behavioral: Engagement-Focused Care Coordination (EFCC)
- Problem Solving Education (PSE) (Active Comparator): The brief Problem Solving Education (PSE) is a six-session cognitive-behavioral program. PSE offers immediate intervention in the PCMH, followed by referral to further treatment if symptoms persist.
  Interventions: Behavioral: Problem Solving Education (PSE)

INTERVENTIONS:
Behavioral: Engagement-Focused Care Coordination (EFCC) — Engagement interviewing is embedded within a traditional PCMH structure using motivational interviewing and shared decision making; it explores treatment options in the context of a patient's life circumstances, and helps her work through ambivalence to receiving care. In one to two sessions, providers disclose the probable diagnosis of depression, provide psycho-education, present treatment options, and engage clients in shared decision making to determine the most appropriate referral.
  Arms: Engagement-Focused Care Coordination (EFCC)
Behavioral: Problem Solving Education (PSE) — Problem solving sessions are one-on-one, workbook-based interactions. Sessions comprise seven sequential steps: 1-defining a problem, 2-establishing goals for problem resolution, 3-generating multiple solution alternatives, 4-Implementing decision making guidelines, 5-evaluating and choosing solutions, 6-Implementing the preferred solutions, and 7-evaluating the outcome.
  Arms: Problem Solving Education (PSE)

SUMMARY:
This is a randomized comparative effectiveness trial to improve outcomes among pregnant and post-partum women with symptoms of depression. Both interventions under study will be based in the patient-centered medical home setting at Boston Medical Center - specifically, in prenatal clinic or in the general pediatrics clinic. The study is a type 1 hybrid effectiveness-implementation trial of 230 mothers with clinically significant depressive symptomatology. Of the 230 subjects, half will receive the Engagement-Focused Care Coordination intervention; the other half will receive the Problem Solving Education intervention. Outcomes for mothers will be assessed every 2 months throughout a 12 month follow-up period. This trial is funded by a contract with PCORI, the Patient-Centered Outcomes Research Institute.

DETAILED DESCRIPTION:
This is a type 1 hybrid effectiveness-implementation trial of 230 mothers with clinically significant depressive symptomatology being conducted at Boston Medical Center (BMC). The effectiveness component of the study (which is the trial registered on ClinicalTrials.gov) is a pragmatic, parallel group randomized trial that measures patient-reported outcomes over 12 months of follow-up. The implementation portion comprises a series of qualitative interviews to discern barriers and facilitators to intervention implementation.

The investigators will enroll 230 mothers with clinically significant depressive symptomatology according to the Edinburgh Postnatal Depression Scale (EPDS), a widely used screening instrument valid during pregnancy and in the postpartum period.

Engagement-Focused Care Coordination will be compared to Problem Solving Education (PSE). Whereas Engagement-Focused Care Coordination emphasizes referral to formal depression services following a brief engagement session, PSE offers initial depression treatment onsite, followed by referral to further care if depressive symptoms persist or worsen. Patients in both arms will have access to the same array of community-based mental health services upon referral. Both intervention arms are designed to be peer-delivered; thus, the investigators will enlist their existing team of PCMH family advocates - a group of women (approximately age-matched with our study participants) - to serve as intervention providers. To minimize contamination across comparators, this team will be divided into those trained in Engagement Interviewing and those trained in PSE.

ELIGIBILITY:
Inclusion Criteria:

* Woman is pregnant and receives prenatal care at BMC; or is biological mother of 0 to 18-month-old child receiving care at BMC pediatric primary care clinic
* Woman has EPDS score ≥ 10
* Woman comfortable speaking and receiving information in English or Spanish
* Woman has no current source of mental health care, defined as having no more than one mental health care appointment in the last 3 months; OR, if more than one appointment, woman has no upcoming appointment

Exclusion Criteria:

* Woman under 18 years of age
* Woman endorses suicidality
* Woman exhibits signs of psychosis or is cognitively limited*

  * As part of the informed consent process, we will administer the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR), which has been validated in populations of depressed and schizophrenic adults

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD MPH, Study Director — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the project study staff will create de-identified datasets and accompanying documentation (data dictionaries, annotated forms and manuals) to be used for data sharing. We will work in collaboration with the Boston University Center for Clinical Translational Epidemiology and Comparative Effectiveness Research, which has a goal of maintaining datasets and collaborating on secondary analyses of clinical trials data.
Supporting Information: Study Protocol, ICF
Time Frame: This will become available approximately one year after the conclusion of the project. We will make the data available indefinitely.
Access Criteria: Access will be determined by the BU Center for Clinical Translational Epidemiology and Comparative Effectiveness Research.

REFERENCES:
- [Derived] Elansary M, Kistin CJ, Antonio J, Fernandez-Pastrana I, Lee-Parritz A, Cabral H, Miller ES, Silverstein M. Effect of Immediate Referral vs a Brief Problem-solving Intervention for Screen-Detected Peripartum Depression: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2313151. doi: 10.1001/jamanetworkopen.2023.13151. PMID 37171819

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 231 were randomized but there was 1 post-randomization exclusion in the PSE group resulting in a sample size of 230 participants.
Period: Allocation
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Started | 115 | 116
Received Allocated Intervention | 88 | 96
Did Not Receive Allocated Intervention | 27 | 19
Completed | 115 | 115
Not Completed | 0 | 1
Not completed — post-randomization exclusion | 0 | 1
Period: Follow-Up
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Started | 115 | 115
Completed | 115 | 114
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Analysis
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Started | 115 | 115
Assessed at 2 Months | 113 | 110
Assessed at 4 Months | 112 | 109
Assessed at 6 Months | 105 | 97
Assessed at 8 Months | 109 | 107
Assessed at 10 Months | 112 | 109
Assessed at 12 Months | 112 | 108
Completed | 115 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE) | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 115 | 115 | 230
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 115 | 230
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 59 | 101
  Not Hispanic or Latino | 73 | 56 | 129
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 21 | 30
  Black | 68 | 57 | 125
  Asian | 2 | 1 | 3
  Other/Multi-race | 23 | 27 | 50
  Missing | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 115 | 115 | 230
Moderate depression based on QIDS score ≥ 11 [Count of Participants; unit: Participants] — Assessed by the Quick Inventory of Depressive Symptoms (QIDS SR-16). This scale is a 16-item self-report measure of depressive symptoms over the past 7 days. Each item is scored 0-3 (0 = no presence of the symptom; 3 = high burden of the symptom), yielding a total score range of 0 to 27. QIDS scores ≥11 suggest moderate depression.
  Participants | 56 | 61 | 117
Anxiety symptoms at baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed by the Beck Anxiety Inventory (BAI).This scale is a 21-item self-report measure of anxiety in the past 7 days. Each item is scored 0-3 (0 = not at all; 3 = severely - it bothered me a lot), yielding a total score range of 0 to 63. The lower the score the less self-reported anxiety.
  score on a scale | 14.9 (11.7) | 15.7 (10.4) | 15.3 (11.05)

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms at 2 Months (QIDS SR-16 ≥ 11)
Description: Assessed by the Quick Inventory of Depressive Symptoms (QIDS SR-16). This scale is a 16-item self-report measure of depressive symptoms over the past 7 days. Each item is scored 0-3 (0 = no presence of the symptom; 3 = high burden of the symptom), yielding a total score range of 0 to 27. QIDS scores ≥11 suggest moderate depression.
Time Frame: 2 months
Population: The overall number of participants analyzed reflects the numbers of participants in each group assessed for this outcome measure time frame as in the participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 113 | 110
Participants | 32 | 26

2. Primary Outcome: Depression Symptoms at 4 Months (QIDS SR-16 ≥ 11)
Description: as for outcome 1
Time Frame: 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
Participants | 29 | 29

3. Primary Outcome: Depression Symptoms at 6 Months (QIDS SR-16 ≥ 11)
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
Participants | 33 | 29

4. Primary Outcome: Depression Symptoms at 8 Months (QIDS SR-16 ≥ 11)
Description: as for outcome 1
Time Frame: 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 109 | 107
Participants | 34 | 33

5. Primary Outcome: Depression Symptoms at 10 Months (QIDS SR-16 ≥ 11)
Description: as for outcome 1
Time Frame: 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
Participants | 30 | 32

6. Primary Outcome: Depression Symptoms at 12 Months (QIDS SR-16 ≥ 11)
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
Participants | 34 | 44

7. Secondary Outcome: Anxiety Symptoms at 2 Months
Description: Assessed by the Beck Anxiety Inventory (BAI).This scale is a 21-item self-report measure of anxiety in the past 7 days. Each item is scored 0-3 (0 = not at all; 3 = severely - it bothered me a lot), yielding a total score range of 0 to 63. The lower the score the less self-reported anxiety.
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 113 | 110
score on a scale | 9.9 (10.2) | 9.4 (8.4)

8. Secondary Outcome: Anxiety Symptoms at 4 Months
Description: as for outcome 7
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
score on a scale | 10.2 (10.3) | 9.9 (9.1)

9. Secondary Outcome: Anxiety Symptoms at 6 Months
Description: as for outcome 7
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
score on a scale | 10.9 (11.0) | 11.4 (10.1)

10. Secondary Outcome: Anxiety Symptoms at 8 Months
Description: as for outcome 7
Time Frame: 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 109 | 107
score on a scale | 10.2 (11.3) | 9.2 (9.7)

11. Secondary Outcome: Anxiety Symptoms at 10 Months
Description: as for outcome 7
Time Frame: 10 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
score on a scale | 9.8 (10.4) | 10.0 (10.5)

12. Secondary Outcome: Anxiety Symptoms at 12 Months
Description: as for outcome 7
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
score on a scale | 10.5 (10.6) | 12.6 (12.2)

13. Secondary Outcome: Engaged With Care at 2 Months
Description: Assessed by the Collaborative Psychiatric Epidemiology Survey (CPES). This 9-item survey records all primary, specialty, and alternative sources of care.
Time Frame: 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 113 | 110
Participants | 15 | 13

14. Secondary Outcome: Engaged With Care at 4 Months
Description: as for outcome 13
Time Frame: 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Engagement-Focused Care Coordination: The brief intervention in Engagement-Focused Care Coordination is the Engagement Interview. In this model, providers meet one to two times with mothers who screen positive for depression, and use techniques of shared decision-making to help mothers process the results of the screen; explore treatment options; and connect with formal mental health services. Engagement-Focused Care Coordination emphasizes referral to formal mental health services.
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
Participants | 19 | 22

15. Secondary Outcome: Engaged With Care at 6 Months
Description: as for outcome 13
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
Participants | 17 | 22

16. Secondary Outcome: Engaged With Care at 8 Months
Description: as for outcome 13
Time Frame: 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 109 | 107
Participants | 17 | 20

17. Secondary Outcome: Engaged With Care at 10 Months
Description: as for outcome 13
Time Frame: 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 109
Participants | 21 | 24

18. Secondary Outcome: Engaged With Care at 12 Months
Description: as for outcome 13
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
Participants | 22 | 26

19. Secondary Outcome: Parenting Behaviors at 6 Months
Description: Assessed by the Parenting Stress Index Short Form (PSI). This 36-item scale yields scores on three subscales - "parental distress", "parent-child dysfunctional interaction", and "difficult child" - which combine to form the total stress scale. Each item is scored 1-5 (1 = strongly agree; 5 = strongly disagree), yielding a scoring range of 36 to 180. Higher scores reflect more parent stress.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
score on a scale | 69.98 (16.53) | 76.93 (18.65)

20. Secondary Outcome: Parenting Behaviors at 12 Months
Description: as for outcome 19
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
score on a scale | 72.92 (16.53) | 79.68 (20.37)

21. Secondary Outcome: Coping With Stress at 6 Months
Description: Assessed by the Problem Focused Subscale of the Brief Coping Orientation to Problems Experienced Inventory (COPE). The overall COPE scale is a 28-item self-report measuring ways of coping with stress. Each item is scored 1-4 (1= I haven't been doing this at all; 4 = I've been doing this a lot). The Problem Focused Subscale includes 6 items focused on active coping, positive reframing, and planning. The scores for each question are added to total the subscale score, which ranges between 6-24 with lower scores indicating less problem-focused coping and higher scores indicating more problem focused coping.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
score on a scale | 13.22 (4.22) | 13.66 (3.94)

22. Secondary Outcome: Coping With Stress at 12 Months
Description: Assessed by the Problem Focused Subscale of the Brief COPE. The overall COPE scale is a 28-item self-report measuring ways of coping with stress. Each item is scored 1-4 (1= I haven't been doing this at all; 4 = I've been doing this a lot). The Problem Focused Subscale includes 6 items focused on active coping, positive reframing, and planning. The scores for each question are added to total the subscale score, which ranges between 6-24 with lower scores indicating less problem-focused coping and higher scores indicating more problem focused coping.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
score on a scale | 12.39 (4.28) | 13.16 (4.18)

23. Secondary Outcome: Behavioral Activation for Depression at 6 Months
Description: Assessed by the Behavioral Activation for Depression Scale (BADS). This 25-item self-reported measure is used to track changes weekly in the behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. The BADS subscales include activation, avoidance/rumination, work/school impairment, and social impairment. Each item is scored 0-6 (0=not at all; 6=completely), yielding a total score range of 0 to 150. High scores indicate greater levels of activation. For all the subscores, high scores are consistent with the subscale name.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination | Problem Solving Education (PSE)
Number analyzed (Participants) | 105 | 97
score on a scale | 93.62 (24.72) | 90.98 (23.70)

24. Secondary Outcome: Behavioral Activation for Depression at 12 Months
Description: as for outcome 23
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
Number analyzed (Participants) | 112 | 108
score on a scale | 95.21 (24.75) | 91.14 (23.27)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Engagement-Focused Care Coordination (EFCC) | Problem Solving Education (PSE)
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115
Other Adverse Events (participants affected / at risk) | 0/115 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03221556/Prot_SAP_000.pdf